CLINICAL TRIAL: NCT01847781
Title: PNEUMOCELL - Conjugated Pneumococcal Vaccination in Patients With Immunoglobulin G-deficiency
Acronym: PNEUMOCELL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Peter Bergman, Associate Professor, Karolinska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2012-004486-41
Record Dates: First submitted 2013-05-01; First posted 2013-05-07 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: IgG Deficiency
Keywords: Opsonophagocytic antibodies; Cellular immunity; Vaccine immunity; Antimicrobial peptides
MeSH Terms: conditions — IgG Deficiency | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IgG-deficient patients (Active Comparator): Prevenar13
  Interventions: Biological: Prevenar13
- Healthy controls (Active Comparator): Prevenar13
  Interventions: Biological: Prevenar13

INTERVENTIONS:
Biological: Prevenar13

SUMMARY:
The aim is to study the immune response to conjugated pneumococcal vaccination (Prevenar13) in Immunoglobulin G-deficient patients and healthy controls. Our hypothesis is that the antibody response will be impaired in patients as compared with controls. In contrast, we postulate that the cellular immune response will be intact.

DETAILED DESCRIPTION:
Ten patients with Immunoglobulin G1 and/or Immunoglobulin G2 deficiency will be enrolled together with 10 age and sex- matched controls. Blood-samples will be drawn at base-line and after 1, 2 and 4 weeks post-vaccination. Serum will be analyzed for opsonophagocytic antibodies. Peripheral blood monocytic cells (PBMCs) will be isolated, frozen and later analyzed for all time-points simultaneously. PBMCs will be stimulated with vaccine-antigens for 3-5 days and cellular activation markers will be measured together with cytokines (Interferon-gamma, Interleukin (IL)-5, IL-13, IL-10, IL-17, IL-22). In addition, levels of antimicrobial peptides in nasal fluid will be measured at baseline and after 4 weeks post-vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Immunoglobulin gamma-deficiency: Immunoglobulin gamma 1-deficiency < 2,8 g/L and/or Immunoglobulin gamma 2-deficiency < 1,15 g/L
* Age 18-65

Exclusion Criteria:

* Immunoglobulin gamma-substitution for 6 months prior to study inclusion
* Prevenar7 or Prevenar13 given prior to study inclusion.
* Pneumovax given during a 2 year period prior to study inclusion
* Pregnancy or planning to become pregnant during the study period (4 weeks)
* Taking part in another clinical study involving drugs or vaccinations during the study period (4 weeks).
* Taking systemic steroids, Non steroidal anti inflammatory drugs (NSAID) or immunosuppressive drugs.
* Being allergic to any substance in the vaccine.
* Acute and ongoing disease with high fever.
* Thrombocytopenia (< 100x109/L).
* Coagulopathy
* Breastfeeding a baby
* The healthy controls should not have any disease with effects on the immune-system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-05; Primary Completion 2013-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in opsonophagocytic antibodies | 4 weeks post-vaccination, change from baseline
  Titers of opsonophagocytic antibodies will be measured at baseline and 4 weeks post-vaccination. Titers from 4 weeks post-vaccination will be compared with baseline-levels.

SECONDARY OUTCOMES:
Change in cellular immunity | 4 weeks post-vaccination, change from baseline
  PBMCs will be collected and stimulated with vaccine-antigens. Cellular activation markers and cytokine release will be measured and results from 4 weeks post-vaccination will be compared with baseline-levels.
Change in antimicrobial peptides | 4 weeks post-vaccination, change from baseline
  Levels of AMPs in nasal fluid will be measured at 0 and 4 weeks post-vaccination. Results from 4 weeks will be compared with base-line levels.

CONTACTS AND LOCATIONS:
Overall Officials: Peter W Bergman, MD, PhD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Immunedeficiency Unit, Karolinska University Hospital, Huddinge, Stockholm, Sweden

REFERENCES:
- [Derived] Zangenah S, Bjorkhem-Bergman L, Norlin AC, Hansen S, Lindqvist L, Henriques-Normark B, Bergman P. The Pneumocell-study: Vaccination of IgG1- and IgG2-deficient patients with Prevnar13. Vaccine. 2017 May 9;35(20):2654-2660. doi: 10.1016/j.vaccine.2017.03.097. Epub 2017 Apr 11. PMID 28410816